CLINICAL TRIAL: NCT01559948
Title: A Randomized Clinical Trial of the Effectiveness of the Compression Belt for Patients With Sacroiliac Joint Pain
Brief Title: Effectiveness of the Compression Belt for Patients With Sacroiliac Joint Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Woman's University (Other)
Collaborators: Texas Physical Therapy Association (Other)
Responsible Party: Principal Investigator, Kelli Brizzolara, Graduate student, Texas Woman's University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16931
Record Dates: First submitted 2012-02-03; First posted 2012-03-21 (Estimated); Results first posted 2019-10-07 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-09

CONDITIONS: Low Back Pain
Keywords: Low back pain; Sacroiliac joint pain; Lumbopelvic stabilization program; Pelvic compression belt; Deep abdominal muscles
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lumbopelvic stabilization exercises plus sacroiliac joint belt (Experimental): The participants will be instructed in the lumbopelvic stabilization program. Additionally, during the initial session, these participants receive a sacroiliac compression belt and be instructed to wear the belt during all waking hours for the first four weeks of the study.
  Interventions: Behavioral: Lumbopelvic stabilization exercise; Device: Sacroiliac joint belt
- Lumbopelvic stabilization exercise (Active Comparator): The participants will be instructed in the lumbopelvic stabilization program.
  Interventions: Behavioral: Lumbopelvic stabilization exercise

INTERVENTIONS:
Behavioral: Lumbopelvic stabilization exercise — The objective of this exercise program is to recruit and train the primary stabilizing muscles of the spine in order for them to more appropriately support the spine. Participants will complete 4 different exercises daily: one in supine, one in standing, one in quadruped, and one in a side-bridge position. The dosage for each exercise is 20 reps with an 8 second hold. In supine, the first exercise is the abdominal drawing-in maneuver. In standing, the first exercise is the abdominal drawing-in maneuver. In quadruped, the first exercise is alternating arm lifts. The final exercise is the side-bridge hold. Participants will then be asked to attend supervised physical therapy sessions twice a week for 2 weeks and once a week for another 2 weeks. They will be instructed to perform the exercises at home daily for a total of 12 weeks as well as complete a compliance log. Progression of the stabilization program will be determined by the physical therapist based on pre-established criteria.
Device: Sacroiliac joint belt — The belt should be worn low around the pelvis just above the greater trochanter and instructed to wear the belt during all waking hours of the first four weeks of the study. The treating physical therapist will monitor the placement of belts during each exercise session. Belt usage logs will be given to each participant to assess compliance with wearing the belt.
  Arms: Lumbopelvic stabilization exercises plus sacroiliac joint belt

SUMMARY:
The purpose of this randomized clinical trial is to examine the usefulness of the addition of a pelvic compression belt to a lumbopelvic stabilization program for patients with sacroiliac joint pain by comparing lumbopelvic stabilization exercises with a pelvic compression belt to lumbopelvic stabilization exercises alone. Outcome measures including the Modified Oswestry Low Back Pain Disability Index (OSW), the percentage change of TrA and IO muscle thickness (i.e. muscle contraction from rest to contract) utilizing ultrasound imaging, the Numeric Pain Rating Scale (NPRS) for pain, and a subjective rating of overall perceived improvement using the Global Rating of Change (GROC) scale will be collected. Hypothesis: The OSW scores and NPRS scores will be lower for those who receive the compression belt in addition to the lumbopelvic stabilization program as compared to those who receive the lumbopelvic stabilization alone. The percent change of muscle thickness for the deep abdominals as well as the GROC scores will be higher for those who receive the compression belt in addition to the lumbopelvic stabilization program as compared to those who receive the lumbopelvic stabilization alone.

DETAILED DESCRIPTION:
Background: The estimated prevalence of sacroiliac joint (SIJ) pain is approximately 13-30% in patients with non-specific low back pain. One common presentation for those with SIJ pain is unilateral pain over the SIJ region, which is described as a positive Fortin's sign. Common impairments for this population include pelvic asymmetry, lumbopelvic muscle imbalance, and decreased lumbopelvic proprioceptive awareness and stability. Two common physical therapy interventions for this population are lumbopelvic stabilization programs and pelvic compression belts. The purpose of this randomized clinical trial is to examine the usefulness of the addition of a pelvic compression belt to a lumbopelvic stabilization program for patients with sacroiliac joint pain by comparing lumbopelvic stabilization exercises with a pelvic compression belt to lumbopelvic stabilization exercises alone. Participants: Thirty participants with unilateral pain near the SIJ will be recruited for the study and randomly assigned to 1 of 2 treatment groups (stabilization plus belt or stabilization alone). Both groups will receive a lumbopelvic stabilization program for 12 weeks. The stabilization plus belt group will also receive a pelvic compression belt to be worn continuously for the first 4 weeks. Outcome measures including the Modified Oswestry Low Back Pain Disability Index (OSW), the percentage change of TrA and IO muscle thickness (i.e. muscle contraction from rest to contract) utilizing ultrasound imaging, the Numeric Pain Rating Scale (NPRS) for pain, and a subjective rating of overall perceived improvement using the Global Rating of Change (GROC) scale will be collected. These outcomes will be assessed at baseline, 4 weeks, and 3 months post-intervention. Hypothesis: The OSW scores and NPRS scores will be lower for those who receive the compression belt in addition to the lumbopelvic stabilization program as compared to those who receive the lumbopelvic stabilization alone. The percent change of muscle thickness for the deep abdominals as well as the GROC scores will be higher for those who receive the compression belt in addition to the lumbopelvic stabilization program as compared to those who receive the lumbopelvic stabilization alone. Data Analysis: Two separate ANOVAs (group x time) with repeated measures will be used to examine the effect of the interventions on disability and the percent change of muscle thickness. Whitney U-test will be used to analyze the NPRS data, and descriptive statistics will be used to report the GROC scores. Clinical Relevance: The results of the study may provide evidence in prescribing pelvic compression belt for those with SIJ pain. It will also offer guidance as to how and when pelvic compression belts should be used in this population. Finally, it will guide physical therapists in prescribing effective interventions for those with SIJ pain.

ELIGIBILITY:
Inclusion Criteria:

* unilateral pain near the sacroiliac joint that does not extend pass the knee
* positive result on 2 of 6 sacroiliac joint provocation tests:

  * compression test
  * distraction test
  * posterior shear test
  * Gaenslens' test (left and right)
  * sacral thrust test

Exclusion Criteria:

* current pregnancy or pregnancy in the last 6 months
* history of surgery to lumbar spine, pelvis, chest, abdomen
* history of congenital lumbar or pelvic anomalies
* any neurological signs in the lower extremity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelli J Brizzolara, MS, Principal Investigator — Texas Woman's University
Locations (1):
- Texas Woman's University, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was a single blinded, mixed-design randomized clinical trial that was conducted in Dallas, Texas from January 2012 to December 2013. Thirty participants with SIJ pain who were not seeking medical care were recruited for this study via flyers and word of mouth marketing.
Pre-assignment Details: Exclusion criteria were current pregnancy or pregnancy in the last six months, history of surgery to the lumbar spine, pelvis, chest, or abdomen, history of congenital lumbar or pelvic anomalies, any neurological signs in the lower extremity, systemic arthritis, and history of pelvic fracture.
Groups:
- Lumbopelvic Stabilization Exc + Belt: The participants will be instructed in the same lumbopelvic stabilization program. Additionally, during the initial session, those participants randomly assigned to the lumbopelvic stabilization plus belt group will also receive a pelvic compression belt.
  Sacroiliac joint belt: Those participants randomly assigned to the lumbopelvic stabilization plus belt group will also receive a pelvic compression belt. They will be taught how to don/doff the belt and instructed to wear the belt during all waking hours for the first 4 weeks of the study. The belt should be worn low around the pelvis just above the greater trochanter. The treating physical therapist will monitor the placement of belts during each exercise session. Belt usage logs will be given to each participant to assess compliance with wearing the belt.
- Lumbopelvic Stabilization Exercise: The participants will be instructed in a lumbopelvic stabilization program.
  Lumbopelvic stabilization exercise: The objective of this exercise program is to recruit and train the primary stabilizing muscles of the spine in order for them to more appropriately support the spine. Participants will then be asked to attend supervised physical therapy sessions twice a week for 2 weeks and once a week for another 2 weeks. They will be instructed to perform the exercises at home daily for a total of 12 weeks as well as complete a compliance log. Progression of the stabilization program will be determined by the physical therapist based on pre-established criteria.
Period: Overall Study
Arm/Group | Lumbopelvic Stabilization Exc + Belt | Lumbopelvic Stabilization Exercise
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Adults, aged 18-65 of any ethnicity with unilateral low back pain that did not extend past the knee with at least two out of 6 positive sacroiliac joint provocation tests.
Groups:
- Lumbopelvic Stabilization Exc + Belt: These participants received a lumbopelvic exercise program plus a pelvic compression belt to wear for the the first four weeks of the study.
- Lumbopelvic Stabilization Exc: The participants received a lumbopelvic exercise program.
- Total: Total of all reporting groups
Arm/Group | Lumbopelvic Stabilization Exc + Belt | Lumbopelvic Stabilization Exc | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.5 (10.6) | 35.5 (12.2) | 31.8 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30
Pain Intensity [Mean (Standard Deviation); unit: units on a scale] — Pain intensity was measured using the Numeric Pain Rating Scale (NPRS). The NPRS is a scale that ranges from 0 (no pain) to 10 (worst pain). Participants were asked to rate their pain intensity on the scale of 0 to 10. A rating of "0" indicated no pain and the higher the number, the worse the pain.
  units on a scale | 3.00 (1.96) | 2.73 (1.34) | 2.9 (1.7)

OUTCOME MEASURES:

1. Primary Outcome: Oswestry Low Back Pain Questionnaire
Description: The Modified Oswestry Back Pain Questionnaire(OSW) will be used to determine Low back pain-related disability. The OSW consists of 10 items assessing different aspects of pain and function related to LBP. Each item is scored 0-5. The item scores are summed and multiplied by 2 to get the total disability score. The total score reported can range from 0-100 with 0 representing no disability and higher scores representing greater disability.
Time Frame: Baseline, 4 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Lumbopelvic Stabilization Exercise Plus Sacroiliac Joint Belt: The participants will be instructed in the same lumbopelvic stabilization program. Additionally, during the initial session, those participants randomly assigned to the lumbopelvic stabilization plus belt group will also receive a pelvic compression belt.
  Sacroiliac joint belt: Those participants randomly assigned to the lumbopelvic stabilization plus belt group will also receive a pelvic compression belt. They will be taught how to don/doff the belt and instructed to wear the belt during all waking hours for the first 4 weeks of the study. The belt should be worn low around the pelvis just above the greater trochanter. The treating physical therapist will monitor the placement of belts during each exercise session. Belt usage logs will be given to each participant to assess compliance with wearing the belt.
Arm/Group | Lumbopelvic Stabilization Exercise Plus Sacroiliac Joint Belt | Lumbopelvic Stabilization Exercise
Number analyzed (Participants) | 15 | 15
units on a scale
  Baseline | 26.00 (10.42) | 24.40 (9.86)
  4 weeks | 17.20 (10.41) | 14.67 (6.49)
  12 weeks | 14.27 (10.08) | 10.00 (8.32)

2. Secondary Outcome: Numeric Pain Rating Scale (NPRS)
Description: The numeric pain rating scale (NPRS) is an 11-point scale with 0 representing "no pain" and 10 representing "worst imaginable pain." This scale will be used to assess pain intensity.
Time Frame: Baseline, 4 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lumbopelvic Stabilization Exc + Belt | Lumbopelvic Stabilization Exercise
Number analyzed (Participants) | 15 | 15
units on a scale
  Baseline | 3.00 (1.96) | 2.73 (1.34)
  4 weeks | 1.20 (1.70) | 1.60 (1.88)
  12 weeks | 1.07 (1.53) | 1.07 (1.58)

3. Secondary Outcome: Percent Change of Muscle Thickness for the Transverse Abdominis (TrA)
Description: The percent change of muscle thickness of the TrA will be assessed using ultrasound imaging. The deep abdominal muscles will be imaged in brightness mode (b-mode) using the SonoSite M-Turbo Ultrasound System. A 2-5 MHz broad spectrum curvilinear transducer will be used to obtain the images. Images were saved for offline analysis using ImageJ software. The muscle thickness for each muscle was determined by the linear distance between the upper and lower fascial lines at the midpoint of the muscle as measured by ImageJ Software. The percent change of muscle thickness was calculated using the following formula: (contracted thickness - resting thickness)/ resting thickness x 100%.
Time Frame: Baseline, 4 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: percentage change
Groups:
- Lumbopelvic Stabilization Exercise Plus Sacroiliac Joint Belt: These participants received a lumbopelvic exercise program plus a pelvic compression belt to wear for the the first four weeks of the study.
- Lumbopelvic Stabilization Excercise: The participants received a lumbopelvic exercise program.
Arm/Group | Lumbopelvic Stabilization Exercise Plus Sacroiliac Joint Belt | Lumbopelvic Stabilization Excercise
Number analyzed (Participants) | 15 | 15
percentage change
  Baseline | 66.52 (21.40) | 81.00 (39.53)
  4 weeks | 141.93 (39.39) | 170.24 (63.95)
  12 weeks | 96.48 (60.44) | 77.02 (40.81)

4. Secondary Outcome: Change in Global Rating of Change (GROC) Scale
Description: The GROC scale will be used to assess the participants' overall perception of improvement since the beginning the interventions. This is a scale ranging from -7 ("a very great deal worse") to 0 ("about the same") to +7 ("a very great deal better").
Time Frame: 4 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Lumbopelvic Stabilization Excercise Plus Sacroiliac Joint Belt: These participants received a lumbopelvic exercise program plus a pelvic compression belt to wear for the the first four weeks of the study.
Arm/Group | Lumbopelvic Stabilization Excercise Plus Sacroiliac Joint Belt | Lumbopelvic Stabilization Excercise
Number analyzed (Participants) | 15 | 15
units on a scale
  4 weeks | 3.13 (2.10) | 3.13 (2.39)
  12 weeks | 4.40 (2.29) | 4.20 (2.21)

5. Secondary Outcome: Percent Change of Muscle Thickness for Internal Oblique
Description: The percent change of muscle thickness of the Internal Oblique will be assessed using ultrasound imaging. The deep abdominal muscles will be imaged in brightness mode (b-mode) using the SonoSite M-Turbo Ultrasound System. A 2-5 MHz broad spectrum curvilinear transducer will be used to obtain the images. Images were saved for offline analysis using ImageJ software. The muscle thickness for was determined by the linear distance between the upper and lower fascial lines at the midpoint of the muscle as measured by ImageJ Software. The percent change of muscle thickness was calculated using the following formula: (contracted thickness - resting thickness)/ resting thickness x 100%.
Time Frame: Baseline, 4 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Lumbopelvic Stabilization Exercise Plus Sacroiliac Joint Belt | Lumbopelvic Stabilization Excercise
Number analyzed (Participants) | 15 | 15
percentage change
  Baseline | 8.23 (11.59) | 5.90 (14.49)
  4 weeks | -21.58 (6.89) | -18.68 (9.59)
  12 weeks | 6.37 (12.34) | 7.65 (14.55)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Lumbopelvic Stabilization Exc + Belt | Lumbopelvic Stabilization Exercise
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No